CLINICAL TRIAL: NCT02192398
Title: Effect of Guanfacine on the Reversal of Opioid-induced Hyperalgesia (OIH)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of NIH funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P-001377; 1R01DA036564-01 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
Keywords: Pain; Pain management; Neck; Back
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia | interventions — Guanfacine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Guanfacine (2mg) (Active Comparator): Subjects will be randomized into 1 of the following 3 treatment groups:
  1. guanfacine (2mg)
  2. guanfacine (1mg)
  3. placebo
  Subjects will be instructed to take one capsule in the evening for 4 weeks.
  Interventions: Drug: Guanfacine
- Guanfacine (1mg) (Active Comparator): Subjects will be randomized into 1 of the following 3 treatment groups:
  1. guanfacine (2mg)
  2. guanfacine (1mg)
  3. placebo
  Subjects will be instructed to take one capsule in the evening for 4 weeks.
  Interventions: Drug: Guanfacine
- Placebo (Placebo Comparator): Subjects will be randomized into 1 of the following 3 treatment groups:
  1. guanfacine (2mg)
  2. guanfacine (1mg)
  3. placebo
  Subjects will be instructed to take one capsule in the evening for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — Subjects will be randomized into 1 of the following 3 treatment groups:
  1. guanfacine (2mg)
  2. guanfacine (1mg)
  3. placebo
  To compare pain threshold, pain tolerance, and wind up, as measured by QST, throughout 4 weeks of drug treatment (guanfacine or placebo).
  Other Names: Tenex, Intuniv
  Arms: Guanfacine (1mg); Guanfacine (2mg)
Drug: Placebo — Subjects will be randomized into 1 of the following 3 treatment groups:
  1. guanfacine (2mg)
  2. guanfacine (1mg)
  3. placebo To compare pain threshold, pain tolerance, and wind up, as measured by QST, throughout 4 weeks of drug treatment (guanfacine or placebo).
  Other Names: Placebo, sugar pill
  Arms: Placebo

SUMMARY:
Combination of guanfacine with opioid medication as a standard treatment for chronic pain.

DETAILED DESCRIPTION:
This aim proposes that guanfacine would be a useful drug to reverse Opioid-Induced Hyperalgesia (OIH) when combined with opioids in chronic pain management.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years old
* Chronic neck or back pain condition for at least 6 months
* VAS score of 4-8, despite opioid therapy
* On a stable morphine equivalent dose of at least 60mg/day and ≤ 240mg/day for at least 3 months

Exclusion Criteria

* Has taken Methadone, Suboxone, Fentanyl, and/or Tramadol in the last six (6) months
* Has taken guanfacine (or other alpha-2AR agonists) in the last six (6) months
* Changes to current or adding new pain treatment while enrolled in the study (i.e. opiates, epidural steroid injection) will be reviewed by the study physician
* Unable to independently provide informed written consent
* Sensory deficits at site of QST, such as peripheral neuropathy
* Intolerable allergies or has had a severe adverse reaction to study medication (i.e. guanfacine, lactose, vitamin B2 a.k.a. riboflavin)
* Takes vitamin B2 > 1.6mg/day during the study
* Pregnant or breastfeeding
* Pending litigation related to neck or back pain
* Diagnosed with Raynaud's syndrome
* Has other chronic pain conditions such as fibromyalgia or joint osteoarthritis that are predominant over back and neck pain with regard to its intensity (VAS)
* Has known pre-existing severe cardiovascular disease (i.e. arrhythmia - prolonged QT interval > 440ms), cerebrovascular disease/accident (i.e., stroke), hepatic or renal impairment, CNS condition, metabolic condition, or history of syncope
* Hypotension (SBP < 90 mmHg and DBP < 60 mmHg for female or SBP < 100 mmHg and DBP < 60 mmHg for male; measured while in a sitting position) will be reviewed by a study physician
* Bradycardia (resting heart rate < 60 bpm) will be reviewed by a study physician
* Subjects are on antihypertensive drugs (e.g., a beta-blocker) that result in hypotension and/or bradycardia as defined above
* Tests positive for illicit drugs, marijuana, or non-prescribed drugs
* Major psychiatric disorders that required hospitalization in the past 6 months such as: major depression, bipolar disorder, schizophrenia, anxiety disorder, or psychotic disorders
* Currently in a treatment program for alcohol or drug abuse, or currently on methadone or buprenorphine (i.e. suboxone, subutex) for treatment of addiction, or currently prescribed stimulants for treatment of ADHD
* History of substance or alcohol abuse (meets DSM IV criteria) per medical record or subject admission
* Subjects are on medications that serve as CYP3A4/5 inhibitors or CYP3A4 inducers including, but are not limited to, valproic acid, macrolide antibiotics, antifungal drugs, St. John wort, ACE inhibitors, nefazodone (antidepressant), calcium channel blockers, H2-receptor antagonists, anti-HIV or AIDS drugs, and antiepileptic drugs
* Subjects are on medications that are ligands for alpha2-adrenergic receptors including antipsychotic drugs (e.g. clozapine) and tricyclic or tetracyclic antidepressants (e.g. imipramine, mirtazapine, mianserin). Any medications taken by a subject at the enrollment will be reviewed regarding their compatibility with guanfacine as well as possible confounding side effects. Subjects will be allowed to take non-opioid pain medications except for gabapentinoids and amitriptyline/nortriptyline as far as such medications do not have incompatibility with guanfacine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | 4 weeks
  Quantitative Sensory Testing (QST) results will be used to compare the 3 treatment groups.

SECONDARY OUTCOMES:
Heat Pain Threshold | 4 weeks
  Subjects will be measured for their heat pain threshold using QST. The testing will be done at 3 of the 4 visits.
Heat Pain Tolerance | 4 weeks
  Subjects will be measured for their heat pain tolerance using QST. The testing will be done at 3 of the 4 visits.
Temporal Pain Summation | 4 weeks
  Subjects will be measured for their temporal pain summation using QST. The testing will be done at 3 of the 4 visits.
Detecting Diffuse Noxious Inhibitory Control (DNIC) | 4 weeks
  Subjects will be measured for their Diffuse Noxious Inhibitory Control (DNIC). The testing will be done at 3 of the 4 visits.
Heat Sensation | 4 weeks
  Subjects will be measured for their heat sensation using QST. The testing will be done at 3 of the 4 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/